CLINICAL TRIAL: NCT05163171
Title: Prevalence of the Victimization and the Perpetration of Intimate Partner Violence Among the Patients From Puy-de-Dôme and Paris Consulting or Being Hospitalized for Addiction Problems and Their Expectations From General Practitioners
Brief Title: Prevalence of the Victimization and the Perpetration of Intimate Partner Violence Among the Patients From Puy-de-Dôme and Paris Consulting or Being Hospitalized for Addiction Problems and Their Expectations From General Practitioners (VIA-MG)
Acronym: VIA-MG
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: General medicine department of Clermont-Ferrand's university (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 VICARD-OLAGNE; 2021-A01356-35 (Other: ANSM)
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Addiction; Violence, Domestic
Keywords: General practice; Intimate partner violence
MeSH Terms: conditions — Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient consulting or hospitalized in addiction structure: patient consulting or hospitalized in addiction structure
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire for conjugal violence prevalence

SUMMARY:
Intimate partner violence and addictions are two frequent problematics with many consequences on health. A link between intimate partner violence and addictions has been found in many studies. Being a drug user increases the risk to be a perpetrator and also a victim of intimate partner violence.

So, it is legitimate to question ourselves about the prevalence of the victims and perpetrators of intimate partner violence among the patients consulting or being hospitalized for an addiction problem. We believe that this prevalence will be high among these patients.

On the other hand, the general practitioners are in first line receiving victims and perpetrators of violence and patients with addiction problems. So it is important to know the profiles of these patients and their expectations from their general practitioners.

DETAILED DESCRIPTION:
The different places where the study will take place are:

* 7 outpatient addiction centers: Addictology consultations in CHU Clermont-Ferrand, CH Sainte-Marie, CH Thiers, CH Ambert, ANPAA (Association Nationale de Prévention en Alcoologie et en Addictologie) of Clermont-Ferrand, Thiers and Ambert.
* 3 hospital addiction centers: Addictology hospital services of CHU of Clermont-Ferrand, CH Thiers and Clémentel.

This study will be based on the filling of self-answered questionnaires by the patients consulting or being hospitalized in the different recruited centers. The questionnaire will be proposed to the patient after the consultation with the practitioner. An information about the study and the anonymity will be given to the patient. The filled questionnaire will be put by the patient in a closed envelope and then in a collection box located in the waiting room.

The different boxes of the different centers will be checked regularly and then the questionnaires will be analysed. The analysis of these questionnaires will allow to describe the population consulting or being hospitalized for addiction problems in the Puy-de-Dôme: age, gender, type of the addiction, the presence of intimate partner violence, associated factors of the violence, recourse characteristics to general practitioners and expectations of GP. We will evaluate the prevalence of victimization and perpetration of intimate partner violence among patients consulting or being hospitalized for addiction problems in the Puy-de-Dôme.

We estimate the duration of the study at around 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18, being or having been in a relationship, consulting or being hospitalized for an addiction problem
* Patient speaking and writing French
* Patient capable of giving his informed consent to take part to the study
* Affiliation to the social security
* Patient who doesn't have a tobacco addiction only

Exclusion Criteria:

* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting or being hospitalized for addiction problems
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of the victimization | day 0
  Prevalence of the victimization and the perpetration of intimate partner violence in patients consulting or being hospitalized for addiction problems who had filled the questionnaire. This prevalence will be measured by the filling of the questions of the self-answered questionnaire by the patients.

SECONDARY OUTCOMES:
Prevalence of each addiction | Day 0
  prevalence will be measured by the filling of the questions of the self-answered questionnaire by the patients.
Socio-demographic characteristics | Day 0
  age in years
Socio-demographic characteristics | Day 0
  male or female
Recourse at general practitioner characteristics | Day 0
  reason and frequency of consultation with their general practitioner
Expectations by the patients of the general practitioners about addictions and intimate partner violence | Day 0
  qualitative answer

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde VICARD-OLAGNE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France